CLINICAL TRIAL: NCT02836535
Title: The Patient-Perspective of Complications After Colon and Rectum Surgery: A Qualitative Analysis
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16-940
Record Dates: First submitted 2016-07-13; First posted 2016-07-19 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2016-08

CONDITIONS: Colorectal Cancer
Keywords: complications; surgery
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- patients with complications: Each subject will participate in an audio-recorded interview, either in-person or by telephone, expected to last 30 to 60 minutes. Subjects' responses to the interview questions and basic demographic data will remain confidential. The interview will examine the impact of complications utilizing a semi-structured script specific to each group
  Interventions: Behavioral: qualitative interviews
- patients without Complications (control group): Each subject will participate in an audio-recorded interview, either in-person or by telephone, expected to last 30 to 60 minutes. Subjects' responses to the interview questions and basic demographic data will remain confidential.
  Interventions: Behavioral: qualitative interviews

INTERVENTIONS:
Behavioral: qualitative interviews

SUMMARY:
The purpose of this study is to understand the patient experience with an adverse event after surgery. An adverse event is an undesirable experience or complication associated with your surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Patients who had elective surgery for a primary colorectal cancer within the last 90 days.
* Patients who either:

  * Develop an eligible complication (Appendix 1) within 30 days of surgery (n = 25 - 30)
  * Do not develop any complication after surgery (n = 25 - 30)

Exclusion Criteria:

* Multivisceral resections
* Metastatic or locally-recurrent disease
* Physical impairment that may prevent participation in an interview or survey setting
* Active psychiatric illness, cognitive or sensory impairment
* Inability to speak or understand English
* Refusal to participate in an audio-recorded interview
* Inability to participate in an audio-recorded interview for reasons not otherwise specified
* Any second surgical procedure unrelated to the complication within the 90-day period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at MSK
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2016-07; Primary Completion 2017-06-28 (Actual); Study Completion 2017-06-28 (Actual)

PRIMARY OUTCOMES:
Number of complications | within 90 days
  Information gathered from these interviews will form the basis for the conceptual model of surgical complications. Qualitative data will be obtained from patients who have directly experienced a surgical complication. These complications are defined and categorized by the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Larissa Temple, MD, MSc, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/